CLINICAL TRIAL: NCT00929461
Title: Do Omega-3 Fatty Acids Have Any Impact On Serum Lactate Levels After Major Gastric Cancer Surgery?
Brief Title: Impact of Omega-3 Fatty Acids on Lactate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Purpose: Treatment
Other Study IDs: B.30.2.EGE.0.01.00.00/7EM/458
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Gastric Surgery
Keywords: omega-3 fatty acids; lactate; surgery; gastric cancer; address the effect of postoperative administration of omega-3 fatty acids on cellular hypoperfusion associated with major gastric surgery.
MeSH Terms: conditions — Stomach Neoplasms | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 group (Other): All patients received TPN for 5 days postoperatively, according to a standard protocol: 3 g/kg BW glucose (5% Dextrose in Ringer's Lactate, Biosel, Istanbul), 1.2 g/kg BW amino acids (Aminosteril 10%, Fresenius-Kabi) and 0.8 g/kg BW omega-6 fatty acids (Lipovenoes® 10%, Fresenius-Kabi) were provided to both groups through an indwelling central venous catheter. In the omega-3 group, the lipid content of TPN was replaced partially by omega-3 fatty acids (Omegaven®, Fresenius-Kabi) up to 0.2 g/kg BW per day.
  Interventions: Drug: Lipovenoes® 10% and Omegaven®,
- Omega 3 + Omega 6 group (Other): All patients received TPN for 5 days postoperatively, according to a standard protocol: 3 g/kg BW glucose (5% Dextrose in Ringer's Lactate, Biosel, Istanbul), 1.2 g/kg BW amino acids (Aminosteril 10%, Fresenius-Kabi) and 0.8 g/kg BW omega-6 fatty acids (Lipovenoes® 10%, Fresenius-Kabi) were provided to both groups through an indwelling central venous catheter.
  Interventions: Drug: Lipovenoes® 10% and Omegaven®,

INTERVENTIONS:
Drug: Lipovenoes® 10% and Omegaven®, — All patients received TPN for 5 days postoperatively, according to a standard protocol: 3 g/kg BW glucose (5% Dextrose in Ringer's Lactate, Biosel, Istanbul), 1.2 g/kg BW amino acids (Aminosteril 10%, Fresenius-Kabi) and 0.8 g/kg BW omega-6 fatty acids (Lipovenoes® 10%, Fresenius-Kabi) were provided to both groups through an indwelling central venous catheter. In the omega-3 group, the lipid content of TPN was replaced partially by omega-3 fatty acids (Omegaven®, Fresenius-Kabi) up to 0.2 g/kg BW per day.

SUMMARY:
Pre- and intra-operative nutritional support in patient undergoing major surgery results in decreased morbidity and mortality. Studies investigating the role of omega-3 fatty acids in these patients are increasing. Some are focused on perfusion at the cellular level. This study was undertaken to address the effect of postoperative administration of omega-3 fatty acids on cellular hypoperfusion associated with major gastric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major gastric cancer surgery

Exclusion Criteria:

* None

Ages: 25 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University General Surgery Dep, Izmir, İzmir, Turkey (Türkiye)

REFERENCES:
- [Result] 16. McNelis J, Marini CP, Jurkiewicz A, et al. Prolonged lactate clearance is associated with increased mortality in the surgical intensive care unit. Am J Surg 2001; 182: 481-5. 7. Smith I, Kumar P, Molloy S, et al. Base excess and lactate as prognostic indicators for patients admitted to intensive care. Intensive Care Med 2001; 27: 74-83. 8. Husain FA, Martin MJ, Mullenix PS, et al. Serum lactate and base deficit as predictors of mortality and morbidity. Am J Surg 2003; 185: 485-91. 9. Skalski M, Goto M, Ravindranath T, et al. Omega-3 polyunsaturated fatty acid enriched diet attenuates stress induced lactacidemia in 10-day-old rats. Pediatr Int 2001; 43: 409-16. 11. Pscheidl EM, Wan JM, Blackburn GL, et al. Influence of omega-3 fatty acids on splanchnic blood flow and lactate metabolism in an endotoxemic rat model. Metabolism 1992; 41: 698-705. 22. Farolan LR, Goto M, Myers TF, et al. Perinatal nutrition enriched with omega-3 polyunsaturated fatty acids attenuates endotoxic shock in newborn rats. Shock 1996; 6: 263-6. 23. Pomposelli JJ, Flores EA, Blackburn GL, et al. Diets enriched with N-3 fatty acids ameliorate lactic acidosis by improving endotoxin-induced tissue hypoperfusion in guinea pigs. Ann Surg 1991; 213:166-76.